CLINICAL TRIAL: NCT03133286
Title: Radiotherapy Assessments During Intervention ANd Treatment (RADIANT)
Acronym: RADIANT
Status: Completed | Type: Observational
Sponsor: DxTerity Diagnostics (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: DXT-RADTOX-AC03; HHSN261201600051C (Other Grant/Funding Number: National Cancer Institute (NCI))
Record Dates: First submitted 2017-04-24; First posted 2017-04-28 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Radiation Therapy; Cancer; Cancer of Anus; Cancer of Bladder; Cancer of Cervix; Cancer of Colon; Cancer of Rectum; Cancer of Esophagus; Cancer of Gallbladder; Cancer of Liver; Cancer of Ovary; Cancer of Pancreas; Cancer of Prostate; Cancer of Kidney and Renal Pelvis; Cancer of Stomach; Cancer of Testis; Cancer of Uterus; Cancer of Uterus and Cervix; Cancer of Kidney
Keywords: Anal Cancer; Bladder; Cervical; Colorectal; Esophageal; Gallbladder; Liver; Ovarian; Pancreas; Pancreatic; Prostate; Rectal; Renal; Kidney; Stomach; Testicular; Uterine; Cancer; Radiation Therapy; Radiation Treatment
MeSH Terms: conditions — Neoplasms; Anus Neoplasms; Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Esophageal Neoplasms; Gallbladder Neoplasms; Liver Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms; Kidney Neoplasms; Stomach Neoplasms; Testicular Neoplasms; Uterine Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Collect blood samples and associated clinical data prior to, during, and post radiation treatment.

DETAILED DESCRIPTION:
In order to further refine and independently validate the performance of DxTerity's test developed during the previous pilot study, the study will collect pre-, during, and post-irradiation blood samples and associated clinical and self-reported information from up to five hundred (500) subjects for analysis. Patients with a diagnosis of primary gastrointestinal (GI), genitourinary (GU), or gynecological (GYN) cancer requiring radiation treatment to the primary disease site will be included in the study. Combining chemotherapy is allowed.

Blood samples for this study will be collected from cancer patients scheduled to undergo radiation therapy prior to and either during or after treatment. Approximately 150μL of blood per time point will be obtained via fingerstick remotely, from the participant's home or doctor's office; participation in this study will not affect any aspect of patient treatment. Samples will be collected using DxTerity's proprietary DxCollect® MCD Fingerstick Kit (MCD).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients age 18 or older
2. Have a permanent address in the United States for the duration of the study
3. Diagnosed with a primary gastrointestinal (GI), genitourinary (GU), or gynecological (GYN) cancer
4. Planned radiation therapy to the abdominal/pelvic area as part of clinical care
5. Able to provide informed consent

Exclusion Criteria:

1. Receipt of radiation within three (3) months to abdominal/pelvic area prior to scheduled start of Radiation Treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients diagnosed with a primary gastrointestinal (GI), genitourinary (GU), or gynecological (GYN) tumors being treated with radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Obtain pre- and post-irradiation participant-collect blood samples | 1.5 years
  Obtain pre-irradiation participant-collected blood sample and associated clinical data from cancer patients undergoing abdominal/pelvic radiation therapy as part of clinical care.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - DxTerity Diagnostics, Compton, California
  - 21st Century Oncology, Bradenton, Florida
  - 21st Century Oncology, Fort Myers, Florida
  - 21st Century Oncology, Plantation, Florida

IPD SHARING:
Plan to Share IPD: No